CLINICAL TRIAL: NCT06517992
Title: Collaborative cOMMUNIty Care for Metastatic breAsT cancEr Patients in inDonesia (Communicated)
Acronym: Communicated
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Collaborators: Pfizer (Industry); Queensland University of Technology (Other)
Responsible Party: Principal Investigator, Martina Sinta Kristanti, Principal Investigator, Gadjah Mada University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Communicated UGM
Record Dates: First submitted 2024-07-11; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Breast Cancer; Cancer
Keywords: Cadre; Education; Community empowerment; Indonesia; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: Quasi experiment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health education for cadre (Experimental): Health education for cadre (Health Community Volunteer) to support metastatic breast cancer patients and their family caregivers
  Interventions: Other: Health education for cadre (communicated project)

INTERVENTIONS:
Other: Health education for cadre (communicated project) — The investigators perform health education to cadre in order to support their role in providing care for metastatic breast cancer living in the community using a module. The module consists of text (written information) and some videos as education medias.

SUMMARY:
The current study aims to empower local cadres in providing care for metastatic breast cancer (mBC) patients in 2 provinces in Indonesia (Bali and Yogyakarta).

DETAILED DESCRIPTION:
Most mBC patients in Indonesia stay at home until they have heavy physical symptoms and need hospitalizations. In this country, even in hospitalization, support from the family caregivers is greatly needed [1]. Family caregivers and the community have a significant role for patients with mBC.

In Indonesia, the support system from local neighbours and community has been implemented for some decades through the involvement of cadres. Health cadres are people from the village who are appointed by their community to train and enhance the community participation in order to empower community health in Indonesia [2]. Most of them are housewives who have enough capability (mentally and physically) to learn, have enough time, and willing to provide support for their community. This role is informal and voluntary-based [3].

-Community support through the existence of cadre in Indonesia- Cadres in Indonesia are initiated by community health services (hereafter Pusat Kesehatan Masyarakat/Puskesmas) around the area. The selection and development of cadres involve the lowest level of local government in the area. Cadres need to have some essential characteristics to undertake their role. They should have empathy as well as good communication skills since one of their tasks is to deliver important health information and message to the community. They need to be able to connect with the community to develop a mutual understanding and be accepted [4]. Funding received from national and local government is allocated for cadres to subsidize the transportation and logistics expenses, but this does not cover the monthly wages [2].

Cadres play a fundamental role in tackling health care problems especially those that are related to psychosocial and cultural factors since they have enough information and knowledge about people and situations in their area. Health care professionals who work in Puskesmas usually cooperate with cadres to gather information related to health conditions in the area or to support local activities. Several roles of cadre have been identified. First, health cadres are responsible for educating and motivating patients and their family to access health care system. They are responsible for assisting patients to access health care facilities for early diagnosis or treatment. On a daily basis, cadres are expected to monitor patients' condition as well as do home visit. At last, it is expected that cadres are able to advocate for patients and their family in the relation to health care professionals [5, 6].

Cadres are initiated and developed by Puskesmas and working closely with integrated health service posts (hereafter Posyandu). Posyandu is a local health unit, under the coordination of Puskesmas, that aims to provide care for baby and infant. Their activities include baby weighting, providing vitamin and enhancing the nutritional status of babies and infants. During Posyandu, health care teams from Puskesmas and cadres are working together. To be able to be classified as active, a Posyandu needs to have at least five health cadres [2]. Currently, there are around 395.495 health cadres in Indonesia.

-Challenges of cadre in Indonesia- In Indonesia, some challenges faced by cadres have been identified. The first is that the role of cadres in Indonesia is still limited. Mostly, their role is merely to provide care for infants and children. Since the number of mBC patients who stay at home is high, health cadres are frequently requested to provide care for this specific group. There have been several initiatives in Indonesia focused on expanding cadres' roles; however, most of the initiatives are focusing on screening and early detection of cancer [7-9]. Until now, there is no single adequate intervention in Indonesia to prepare cadres in Indonesia to support mBC patients and their family caregivers.

The second issue is that although cadres have some connections with Puskesmas, the breadth and depth of the connections are still limited and have an unclear structure. There is a need to open communication channels so that cadres are able to connect with health care professionals from Puskesmas and their role can be recognized by local health authorities. When needed, cadres would be better positioned to request for help or provide important information to Puskesmas in regards to mBC patients problems and needs.

Given the important role of cadres, the COMMUNICATED project aims to empower local cadres to provide care for metastatic breast cancer (mBC) patients in in Indonesia.

ELIGIBILITY:
Inclusion Criteria for mBC:

* Diagnosed for having breast cancer at least in stage 3B or confirm to have metastatic breast cancer
* Live at home
* Considered as adult (Eighteen years of age or older)

Exclusion Criteria for mBC:

- mBC patients will be exclude when their physical condition is deteriorating or when they need hospitalization.

The following criteria will be applied for family caregivers:

1. Appointed by mBC patients or self-identified as family caregiver of mBC patients for at least 3 months
2. Live/not live together with mBC patients but providing care to mBC patient
3. Considered as adult (Eighteen years of age or older)

Inclusion criteria for cadre:

The local cadre in Yogyakarta and Bali who self-identified as local cadre in the community and willing to involve for assisting mBC patients. The local cadre will be excluded when they are not providing consent to involve in the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female metastatic Breast cancer
Enrollment: 80 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
European Organization for Research and Treatment for Cancer Quality of Life Questionnaire - Breast Cancer (EORTC QLQ-BR23) | 2-3 months
  Questionnaire to measure Quality of Life of Breast Cancer Patients. This consists of 23 items with 2 domains: symptom scales (systemic therapy side effects, upset by hair loss, Arm symptoms and Breast symptoms) and functional scale (body image, future perspective, sexual functioning, and sexual enjoyment). The questionnaire uses likert scale 1-4. The options are not at all, a little, quite a bit, and very much. An option for "Not applicable (N/A)" is also offered for an item of sexual enjoyment. This instrument has been translated to Bahasa Indonesia. The scale ranges in score from 0-100 with a higher score for the functional scale represents a high or healthy level of functioning. On the other hand, the high score for symptom scale represents frequent problems.

SECONDARY OUTCOMES:
Symptom Management Self Efficacy Scale - Breast Cancer (SMSES-BC) | 2-3 months
  This instrument consists of 27 items related to self-efficacy in the symptom management relevant to chemotherapy for patients with breast cancer. The items is offering rating from 0 not at all confident) to 10 (completely confident). The higher score represents higher perceived of symptom-management self-efficacy.
Preparedness for caregiving scale (PCS) | 2-3 months
  PCS consists of 8 items and 1 open ended question. This is a family caregiver instrument to self-rated how well are of becoming caregivers with the domain of providing physical care, emotional support, setting up in-home support services and dealing with caregiver's stress. Responses are ranging from 0 (not at all prepared) to 5 (very well prepared).
Resilience Scale Specific to Cancer (RS-SC-10) | 2-3 months
  tThis instrument is a brief and validated instrument for family caregivers of patient with cancer [44] which consists of 10 items. RS-SC developed using MRIT analysis and consists of 2 domains: generic and Shift-Persist. The score ranges from 10-50 with the higher score represents higher resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Syahirul Alim, PhD, Study Chair — Faculty of Medicine, Public Health and Nursing, Universitas Gadjah Mada
Locations (2):
- Indonesia (2):
  - Primary Health Center, Yogyakarta, Special Region of Yogyakarta
  - Primary Health center, Bali

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kristanti MS, Effendy C, Utarini A, Vernooij-Dassen M, Engels Y. The experience of family caregivers of patients with cancer in an Asian country: A grounded theory approach. Palliat Med. 2019 Jun;33(6):676-684. doi: 10.1177/0269216319833260. Epub 2019 Mar 27. PMID 30916614
- [Result] Kristanti MS, Setiyarini S, Effendy C. Enhancing the quality of life for palliative care cancer patients in Indonesia through family caregivers: a pilot study of basic skills training. BMC Palliat Care. 2017 Jan 17;16(1):4. doi: 10.1186/s12904-016-0178-4. PMID 28095837
- See also: Sapar, Salju, Risal M, et al. The influence of TB care community cadre's roles on the treatment adherence of tuberculosis (TB) sufferers. Enfermería Clínica 2020; 30: 244-248. — https://doi.org/10.1016/j.enfcli.2020.06.056
- See also: Sunarti. peran kader kesehatan dalam pelayanan posyandu UPTD puskesmas kecamatan sananwetan kota Blitar. Jurnal Keperawatan Malang 2019; 3: 94-100. — https://jurnal.stikespantiwaluya.ac.id/index.php/JPW/article/view/63